CLINICAL TRIAL: NCT04717765
Title: Photobiomodulation With Low Level Laser in the Prevention and Treatment of Oral Lesions (Mucositis, Hyposalivation and Osteonecrosis) Resulting From Anti-neoplastic Treatment With Chemotherapy or Radiotherapy.
Brief Title: Photobiomodulation in Oral Lesions Resulting From Anti-neoplastic Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Mario Pérez Sayáns, Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCT-LB-VE-20
Record Dates: First submitted 2021-01-11; First posted 2021-01-22 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Oral Mucositis; Osteoradionecrosis; Osteonecroses, Bisphosphonate; Osteonecrosis Due to Drugs, Jaw; Hyposalivation; Head and Neck Cancer; Oral Cancer
Keywords: Dentistry; Health Promotion; Clinical trial; Oral Mucositis; Radiotherapy; Chemotherapy; Lasertherapy; Phototherapy; Hyposalivation; ORN; MRONJ
MeSH Terms: conditions — Stomatitis; Osteoradionecrosis; Bisphosphonate-Associated Osteonecrosis of the Jaw; Xerostomia; Head and Neck Neoplasms; Mouth Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Preventive in oral mucositis caused by chemo or radiotherapy - LLL Phototherapy (Experimental): Application of LLL phototherapy from the first day until the last day, on all days that the chemo or radiotherapy treatment is administered. If the patient still shows evidence of mucositis at the end of the treatment, additional applications can be performed.
  Application: in wavelength 660 nm (red), there will be 78 intra oral points, with a time of 10 seconds per point, at a power of 100 mw, totaling a power of 1J per point.
  Interventions: Device: Preventive, LLL Phototherapy and topical Vit E
- Preventive in oral mucositis caused by chemo or radiotherapy - Vit E (Active Comparator): Topical Vit. E spray, from the first day to the last day, every day that the chemo or radiotherapy treatment is administered.
  Application: on the first day the professional will demonstrate the application on intra-oral mucous points. On the other days the patient will do self application, twice a day.
  Interventions: Device: Preventive, LLL Phototherapy and topical Vit E
- Preventive in oral mucositis caused by chemo or radiotherapy - mouthwash (No Intervention): Oral hygiene control and mouthwash with chlorhexidine 0.12%, from the first to the last day of administration of the chemo or radiotherapy treatment. On the first day the professional will demonstrate the care. On the other days the care will be taken by the patient himself, for at least three times a day.
- Curative in oral mucositis caused by chemo or radiotherapy - LLL Phototherapy (Experimental): Application of LLL phototherapy from the tenth day until the last day, on all days that the chemo or radiotherapy treatment is administered. If the patient still shows evidence of mucositis at the end of the treatment, additional applications can be performed.
  Application: in wavelength 660 nm (red), there will be 78 intra oral points, with a time of 10 seconds per point, at a power of 100 mw, totaling a power of 1J per point.
  Interventions: Device: Curative, LLL Phototherapy and topical Vit E
- Curative in oral mucositis caused by chemo or radiotherapy - mucositis Vit E (Active Comparator): Topical Vit. E spray, application from the tenth day, and until the last day, every day that the chemo or radiotherapy treatment is administered.
  Application: on the first day the professional will demonstrate the application on intra-oral mucous points. On the other days the patient will do self application, twice a day.
  Interventions: Device: Curative, LLL Phototherapy and topical Vit E
- Curative in oral mucositis caused by chemo or radiotherapy- mouthwash (No Intervention): Oral hygiene control and mouthwash with chlorhexidine 0.12%, from the tenth to the last day of administration of the chemo or radiotherapy treatment. On the first day the professional will demonstrate the care. On the other days the care will be taken by the patient himself, for at least three times a day.
- Preventive osteonecrosis resulting from chemo or radiotherapy - LLL Phototherapy + extraction (Experimental): For patients who need dental extraction for the adequacy of the oral cavity. Application of LLL phototherapy on the day the dental extraction is performed and every 72hr, totaling 5 applications. It must be done at least 3 months before the beginning of the chemo or radiotherapy treatment.
  Application: in wavelength 660 nm (red), alveolar ridge, 1 point per cm², with a time of 10 seconds per point, at a power of 100 mw, totaling a power of 1J per point. In wavelength 808 nm (infrared), buccal and lingual/palatal board 2 points in the length of the root, with a time of 20 seconds per point, at a power of 100 mw, totaling a power of 2J per point.
  Interventions: Device: Preventive, LLL Phototherapy and LPRF
- Preventive osteonecrosis resulting from chemo or radiotherapy - LPRF+ extraction (Active Comparator): For patients who need dental extraction for the adequacy of the oral cavity. LPRF placement on the day the tooth extraction is performed. The procedure must be performed at least 3 months before the start of chemo or radiotherapy treatment.
  After the LPRF has been placed, the suture should be done in a way that facilitates healing for primary intention.
  Interventions: Device: Preventive, LLL Phototherapy and LPRF
- Preventive osteonecrosis resulting from chemo or radiotherapy - extraction only (No Intervention): For patients who need dental extraction for the adequacy of the oral cavity, the procedure must be performed at least 3 months before the start of chemo or radiotherapy treatment.
  The suture should be done in a way that facilitates healing for primary intention.
- Curative osteonecrosis resulting from chemo or radiotherapy - LLL Phototherapy + sequestrectomy (Experimental): Patients who have been diagnosed with bone necrosis after treatment with chemo or radiotherapy, clinical confirmation and radiography. Bone sequestrectomy, removal of necrotic tissue and application of LLL phototherapy on the day of surgery and every 72hr, totaling 5 applications. The suture should be done in a way to facilitate healing for primary intention.
  Application: in wavelength 660 nm (red), alveolar ridge, 1 point per cm², with a time of 10 seconds per point, at a power of 100 mw, totaling a power of 1J per point. In wavelength 808 nm (infrared), buccal and lingual/palatal board 2 points in the length of what would be the dental root, with a time of 20 seconds per point, at a power of 100 mw, totaling a power of 2J per point.
  Interventions: Device: Curative, LLL Phototherapy and LPRF
- Curative osteonecrosis resulting from chemo or radiotherapy - LPRF + sequestrectomy (Active Comparator): Patients who have been diagnosed with bone necrosis after treatment with chemo or radiotherapy, clinical confirmation and radiography. Bone sequestrectomy, removal of necrotic tissue and placement of the LPRF on the day of surgery will be performed.
  After the LPRF is placed, the suture should be done in a way that facilitates healing for primary intention.
  Interventions: Device: Curative, LLL Phototherapy and LPRF
- Curative osteonecrosis resulting from chemo or radiotherapy - sequestrectomy only (No Intervention): Patients who were diagnosed with bone necrosis after treatment with chemo or radiotherapy, clinical confirmation and radiography. Bone sequestrectomy and removal of necrotic tissue will be performed.
  The suture should be done in a way that facilitates healing for primary intention.

INTERVENTIONS:
Device: Preventive, LLL Phototherapy and topical Vit E — Interventions will be carried out for patients who have already passed or will undergo anti-neoplastic chemotherapy or radiation therapy.
  Arms: Preventive in oral mucositis caused by chemo or radiotherapy - LLL Phototherapy; Preventive in oral mucositis caused by chemo or radiotherapy - Vit E
Device: Curative, LLL Phototherapy and topical Vit E — Interventions will be carried out for patients who have already passed or will undergo anti-neoplastic chemotherapy or radiation therapy.
  Arms: Curative in oral mucositis caused by chemo or radiotherapy - LLL Phototherapy; Curative in oral mucositis caused by chemo or radiotherapy - mucositis Vit E
Device: Preventive, LLL Phototherapy and LPRF — Interventions will be carried out for patients who have already passed or will undergo anti-neoplastic chemotherapy or radiation therapy.
  Arms: Preventive osteonecrosis resulting from chemo or radiotherapy - LLL Phototherapy + extraction; Preventive osteonecrosis resulting from chemo or radiotherapy - LPRF+ extraction
Device: Curative, LLL Phototherapy and LPRF — Interventions will be carried out for patients who have already passed or will undergo anti-neoplastic chemotherapy or radiation therapy.
  Arms: Curative osteonecrosis resulting from chemo or radiotherapy - LLL Phototherapy + sequestrectomy; Curative osteonecrosis resulting from chemo or radiotherapy - LPRF + sequestrectomy

SUMMARY:
Introduction: There are several manifestations in the oral mucosa resulting from antineoplastic treatments by chemo (QT) or radiotherapy (RT). In this study we will collect the variables referring to oral mucositis (OM), radiodermatitis, osteonecrosis of the jaws (ONJ), hyposalivation and xerostomia, dysgeusia, pain, oral candidiasis (opportunistic infection), trismus, quality of life, oral hygiene.

MO and hyposalivation, which are related to damage to the salivary glands, are the most common manifestations, and ONJ is the most difficult to treat. The dentist can play an important role in prevention and treatment these oral lesions, directly influencing the patient's quality of life and adherence to antineoplastic treatment.

Objectives: The main objective is to evaluate the efficacy of the intervention, using LLL phototherapy and topical Vit E, in the OM. And the intervention through LLL phototherapy and LPRP in the ONJ. These interventions will be performed by dentists during antineoplastic medical treatment.

Material and methods: clinical trial, randomized, with balanced randomization, single-blind (for the evaluator of the results) with 2 experimental arms and a control group, carried out in a single center. Group 1, intervention with LLL phototherapy, Group 2, intervention with application of topical Vit E and Group 3, mouthwash with 0.12% chlorhexidine (usual clinical information). 360 patients will participate in this study from the Units of Oncology Medicine, Radiotetaphic Medicine and Oral Medicine, Oral Surgery and Implantology at the University of Santiago de Compostela. The segment of the patients will be given, an initial visit and returns every day that hears the application of antineoplastic treatment for the group of LLL phototherapy, returns of 15 days, one month, three months, six months, nine months and one year. In these return visits, evaluations and questionnaires will be carried out regarding all the variables that we will collect.

Predictable results: If the application of laser phototherapy or topical Vit E contributes to the cessation, reduction or improvement of the clinical evolution of the manifestation of oral lesions, these treatments could be immediately implemented in our Oral Medicine unit and could lay the foundations for its implementation in different public centers and private.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck or breast cancer who will undergo chemotherapy or radiotherapy.

Exclusion Criteria:

* Participants who do not sign the informed consent.
* Patients who have been or will be treated by chemo and radiotherapy together.
* Patients in treatment of a cancer recurrence.
* Patients reporting diabetes or sjogren's syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Prevention of oral mucositis with LLL phototherapy, evaluation using NCI-CTC mucositis scale of the "National Cancer Institute" - grade 1 to 5 - Chemotherapy | 3 months
  The main objective is to evaluate whether LLL phototherapy acts on preventing oral mucositis in patients who will receive chemotherapy. The result will be determined by the percentage of patients who reduce the intensity of the manifestation and/or do not develop oral mucositis, for this we will use the NCI-CTC mucositis scale of the "National Cancer Institute". Grade refers to the severity. Grades 1 through 5 (the most severe).
  Will be compared to those who receive topical Vit. E or chlorhexidine mouthwash, in the prevention arms of the study.
Prevention of osteonecrosis of the jaws with LLL phototherapy, evaluation using the MASCC scale - stage 1 to 3 - Chemotherapy | 6 months
  The main objective is to assess whether LLL phototherapy works to prevent bone necrosis of the jaws in patients who need dental extractions and who will still receive chemotherapy. The result will be determined by the percentage of patients who do not develop bone necrosis after extraction and phototherapy, the " Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO/ASCO) Clinical Practice Guideline on Medication-Related Osteonecrosis of the Jaw" will be used for classification of bone necroses. Stage refers to the severity. Stages 1 through 3 (the most severe).
  It will be compared with those who receive LPRF after extraction or only extraction, in the prevention arms of the study.
Treatment of oral mucositis with LLL phototherapy, evaluation using NCI-CTC mucositis scale of the "National Cancer Institute" - grade 1 to 5 - Chemotherapy | 3 months
  The main objective is to evaluate the efficacy of LLL phototherapy in the LLL phototherapy treating. The result will be determined by percentage of patients who develop oral mucositis after the first 10 days of treatment with chemotherapy, and who receive phototherapy, and have rapid regression of oral mucositis, for this we will use the NCI-CTC mucositis scale of the "National Cancer Institute". Grade refers to the severity. Grades 1 through 5 (the most severe).
  Will be compared with patients receiving topical Vit. E or chlorhexidine mouthwash.
Treatment of osteonecrosis of the jaws with LLL phototherapy, evaluation using the MASCC scale - stage 1 to 3 - Chemotherapy | 6 months
  The main objective is to evaluate the efficacy of LLL phototherapy in the treatment of osteonecrosis of the jaws in patients with bone necrosis after receiving chemotherapy. The result will be determined by the percentage of patients who are cured of osteonecrosis after sequestromia and phototherapy, for this which we will use the " Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO/ASCO) Clinical Practice Guideline on Medication-Related Osteonecrosis of the Jaw" will be used for classification of bone necroses. Stage refers to the severity. Stages 1 through 3 (the most severe).
  It will be compared to those who receive sequestromia and LPRF or just sequestromia.
Prevention of oral mucositis with LLL phototherapy, evaluation using NCI-CTC mucositis scale of the "National Cancer Institute" - grade 1 to 5 - Radiotherapy | 3 months
  The main objective is to evaluate whether LLL phototherapy acts on preventing oral mucositis in patients who will receive radiotherapy. The result will be determined by the percentage of patients who reduce the intensity of the manifestation and/or do not develop oral mucositis, for this we will use the NCI-CTC mucositis scale of the "National Cancer Institute". Grade refers to the severity. Grades 1 through 5 (the most severe).
  Will be compared with patients receiving topical Vit. E or chlorhexidine mouthwash.
Prevention of osteonecrosis of the jaws with LLL phototherapy, evaluation using Notani scale - grade 1 to 3 - Radiotherapy | 6 months
  The main objective is to assess whether LLL phototherapy works to prevent bone necrosis of the jaws in patients who need dental extractions and who will still receive radiotherapy. The result will be determined by the percentage of patients who do not develop bone necrosis after extraction and phototherapy, the Notani scale, will be used for classification of bone necroses. Grade refers to the severity. Grades 1 through 3 (the most severe).
Treatment of oral mucositis with LLL phototherapy, evaluation using NCI-CTC mucositis scale of the "National Cancer Institute" - grade 1 to 5 - Radiotherapy | 3 months
  The main objective is to evaluate the efficacy of LLL phototherapy in the LLL phototherapy treating. The result will be determined by percentage of patients who develop oral mucositis after the first 10 days of treatment with radiotherapy, and who receive phototherapy, and have rapid regression of oral mucositis, for this we will use the NCI-CTC mucositis scale of the "National Cancer Institute". Grade refers to the severity. Grades 1 through 5 (the most severe).
  Will be compared with patients receiving topical Vit. E or chlorhexidine mouthwash.
Treatment of osteonecrosis of the jaws with LLL phototherapy, evaluation using Notani scale - grade 1 to 3 - Radiotherapy | 6 months
  The main objective is to evaluate the efficacy of LLL phototherapy in the treatment of osteonecrosis of the jaws in patients with bone necrosis after receiving radiotherapy. The result will be determined by the percentage of patients who are cured of osteonecrosis after sequestromia and phototherapy, for which we will use the Notoni Scale. Grade refers to the severity. Grades 1 through 3 (the most severe).

SECONDARY OUTCOMES:
Interference of oral mucositis with quality of life - QLQ-C30 test | 6 months
  The quality of life of all patients in the mucositis study, whether chemotherapy or radiotherapy, preventive or curative, will be estimated using the EORTC core Quality of Life questionnaire QLQ-C30.
Interference of osteonecrosis of the jaws with quality of life - QLQ-C30 test | 12 months
  The quality of life of all patients in the mucositis study, whether chemotherapy or radiotherapy, preventive or curative, will be estimated using the EORTC core Quality of Life questionnaire QLQ-C30.
Hyposalivation with global saliva test - Oral mucositis | 6 months
  Alteration of salivary glands will be estimated by measurement; hyposalivation, by global saliva test, stimulated and unstimulated saliva, (GST l and ll).
  Rates of less than 0.1-0.2ml/min for resting saliva and less than 0.5-0.7ml/min for stimulated saliva are considered abnormal.
Xerostomia with s will be estimated by measurement. Xerostomia, with Xerostomia inventory - Oral mucositis | 6 months
  Alteration of salivary glands will be estimated by measurement. Xerostomia, by "Xerostomia inventory" a questionnaire containing 11 questions, with the intention of measure a subjective sensation of the patient.
Pain assessed by EVA - score 0 to 10 - all patients | 6 months
  Pain will also be measured in all groups of the study, through the visual analogue - EVA Scale, adapted for pain.
  Subjective evaluation of pain, indicated by the patient. Scale from 0 to 10 (the most intense).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico Universitário, Santiago de Compostela, LA Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We will anonymize and categorize the clinical data of the patients to share the information with the other researchers of the group.